CLINICAL TRIAL: NCT01472614
Title: Effect of Add-on Therapy With DLBS3233 on Glycemic Control, Lipid Profile, and Adiponectin in Patients With Type-2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Add-on Therapy With DLBS3233 in Patients With Type-2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLBS3233-0411
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Type-2 Diabetes Mellitus
Keywords: Type-2 diabetes mellitus; Add-on therapy
MeSH Terms: interventions — DLBS3233

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLBS3233 (Experimental)
  Interventions: Drug: DLBS3233

INTERVENTIONS:
Drug: DLBS3233 — Study treatment will be DLBS3233 at a dose of 100 mg once daily (for 12 weeks) in addition to current anti-diabetic treatment used by respective study subjects and treatment intensification (lifestyle modification)
  Other Names: Inlacin

SUMMARY:
This is an open clinical study for 12 weeks of therapy to investigate clinical efficacy and safety of an add-on therapy with DLBS3233 in improving blood glucose control, lipid profile, and adiponectin in subjects with type-2 diabetes mellitus.

DETAILED DESCRIPTION:
There will only be one group in this study who will receive study treatment as follows: anti-diabetic agents currently used by respective subjects for at least 3 months prior to Screening, treatment intensification (lifestyle modification), and DLBS3233 at a dose of 100 mg once daily for 12 weeks.

Clinical and laboratory examinations to evaluate the investigational drug's efficacy and safety will be performed at baseline and at interval of 6 weeks over the 12-week course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with age of 40 - 70 years; or female subjects with age of 55 - 70 years (post-menopause) at screening
* Diagnosed with type-2 diabetes mellitus
* Have been being treated with a combination of two OHA for at least 3 months prior to screening
* A1c level of >= 7.0 %
* Hemoglobin level of >= 10 g/dL
* Body Mass Index (BMI) > 18.5 kg/m2
* Refuse insulin therapy
* Able to take oral medicine

Exclusion Criteria:

* Subjects with symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Uncontrolled hypertension defined as systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
* History of or current chronic treatment with insulin
* History of renal and/or liver disease
* Impaired liver function: serum ALT > 2.5 times upper limit of normal and positive result of chronic or acute hepatitis B or C test
* Impaired renal function: serum creatinine >= 1.5 times upper limit of normal
* Current treatment with systemic corticosteroids or herbal (alternative) medicines
* Any other disease state or uncontrolled illness, which judged by the investigator, could interfere with trial participation or trial evaluation
* Participation in any other clinical studies within 30 days prior to screening

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduction of A1c level | 12 weeks
  Reduction of A1c level from baseline after 12 weeks of treatment

SECONDARY OUTCOMES:
Reduction of venous A1c level | 6 weeks
  Reduction of venous A1c level from baseline to 6 weeks of treatment
Reduction of venous FPG | 6 and 12 weeks
  Reduction of venous FPG from baseline to every evaluation-time point
Reduction of venous 1h-PG | 6 and 12 weeks
  Reduction of venous 1 hour-post prandial plasma glucose from baseline to every evaluation-time point
Change in fasting insulin level | 6 and 12 weeks
  Change in fasting insulin level from baseline to every evaluation-time point
Change in HOMA-R | 6 and 12 weeks
  Change in HOMA-R from baseline to every evaluation-time point
Change in HOMA-B | 6 and 12 weeks
  Change in HOMA-B from baseline to every evaluation-time point
Change in adiponectin level | 6 and 12 weeks
  Change in adiponectin level from baseline to every evaluation-time point
Change in lipid profile | 6 and 12 weeks
  Change in lipid profile from baseline to every evaluation-time point, including: LDL-cholesterol (direct), HDL-cholesterol, total cholesterol, and triglycerides
Change in body weight | 6 and 12 weeks
  Change in body weight from baseline to every evaluation-time point
Hematology | 6 and 12 weeks
  Hematology parameters (Hemoglobin level, Hematocrit, Red Blood Cell count, White Blood Cell count as well as its differentials, and platelet count) will be evaluated at baseline, at interval of 6 weeks, and at the end of study
Liver function | 6 and 12 weeks
  Liver function parameters (serum ALT, serum AST, gamma-glutamyl transferase, alkaline phosphatase, and total bilirubin levels) will be measured at baseline, at interval of 6 weeks, and at the end of study
Renal function | 6 and 12 weeks
  Renal function parameter, i.e. serum creatinine level will be measured at baseline, at interval of 6 weeks, and at the end of study
Adverse events | 1-12 weeks
  Adverse events as well as number of subjects experienced the events will be observed and evaluated during the study period (12 weeks) and until all adverse events have been recovered or stabilized.

CONTACTS AND LOCATIONS:
Overall Officials: Askandar Tjokroprawiro, Prof.Dr.dr,SpPD-KEMD,FINASIM, Principal Investigator — Surabaya Diabetes and Nutrition Center, Dr. Soetomo Hospital
Locations (2):
- Indonesia (2):
  - Private Clinic at Jl. Prof. Dr. Moestopo 164, Surabaya, East Java
  - Surabaya Diabetes and Nutrition Centre, Dr. Soetomo Hospital, Surabaya, East Java